CLINICAL TRIAL: NCT02745730
Title: Resting State Functional Magnetic Resonance Imaging of Human Brain Responses to Nutrient Shake
Brief Title: RS-fMRI to Nutrient Shakes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: REF-ICE-2421
Record Dates: First submitted 2016-04-04; First posted 2016-04-20 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Pleasure
MeSH Terms: interventions — Glucose; Fructose; trichlorosucrose; psicose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Glucose (Active Comparator): Shake sweetened with glucose
  Interventions: Other: Glucose
- Fructose (Active Comparator): Shake sweetened with fructose
  Interventions: Other: Fructose
- Sucralose (Experimental): Shake sweetened with sucralose
  Interventions: Other: Sucralose
- Allulose (Experimental): Shake sweetened with allulose
  Interventions: Other: Allulose

INTERVENTIONS:
Other: Glucose
  Arms: Glucose
Other: Fructose
  Arms: Fructose
Other: Sucralose
  Arms: Sucralose
Other: Allulose
  Arms: Allulose

SUMMARY:
Resting state functional magnetic resonance imaging (rsfMRl) of the brain is used to measure pleasantness after consumption of four different milkshakes with added sugars or sweeteners.

DETAILED DESCRIPTION:
The central role of the brain in regulating food intake and steering feeding behaviour is increasingly recognized. It is currently well accepted that the brain is the target organ to measure the effects of pleasantness and energy homeostasis in order to change feeding behaviour to reduce the rising prevalence of obesity. The effects of food on the brain are multiple and complex. In addition to primary aspects of food such as taste, texture, looks and smell, secondary aspects such as energy regulation are as much important in the entire "eating experience". Resting state functional connectivity in the brain can be assessed by the analysis of low-frequency fluctuations present in the blood-oxygenation-level-dependent (BOLD) signal in functional magnetic resonance imaging (fMRI). Investigators will use resting state functional magnetic resonance imaging (rsfMRl) to detect changes in connectivity in the default mode and salience network after consumption of four different milkshakes with added sugars or sweeteners.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age between 18 and 25 years
* BMI between 20 and 23 kg/m2
* Weight above 70 kg
* Length between 170 and 190 centimetres

Exclusion Criteria:

* Diabetes or history of other disturbances of glucose metabolism (eg impaired glucose tolerance, hypoglycaemia).
* Any genetic or psychiatric disease (e.g. fragile X syndrome, major depression) affecting brain
* Any know food allergy or intolerance
* Any significant chronic disease
* Renal or hepatic disease
* Recent weight changes or attempts to lose weight (> 3 kg weight gain or loss, within the last 3 months)
* Smoking (current or last 6 months)
* Alcohol consumption of more than 21 units per week or use of recreational drugs at present or in the last year
* Recent blood donation (within the last 2 months)
* Recent participation in other biomedical research projects (within the last 3 months), participation in 3 or more biomedical research projects in one year
* Contra-indication to MRI scanning:

  * Claustrophobia
  * Pacemakers and defibrillators
  * Nerve stimulators
  * Intracranial clips
  * intraorbital or intraocular metallic fragments
  * Cochlear implants
  * Ferromagnetic implants

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03; Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the connectivity in the default mode and salience network: glucose and fructose vs. sucralose and allulose. | Six minutes before (baseline) and 12 minutes after (response) test product intake

SECONDARY OUTCOMES:
2. Change from baseline in the connectivity in the default mode and salience network: glucose vs. fructose. | Six minutes before (baseline) and 12 minutes after (response) test product intake
3. Change from baseline in the connectivity in the default mode and salience network: allulose vs. sucralose. | Six minutes before (baseline) and 12 minutes after (response) test product intake

OTHER OUTCOMES:
4. Change from baseline in the connectivity in the default mode and salience network: glucose vs allulose; glucose vs sucralose; fructose vs sucralose and fructose vs allulose. | Six minutes before (baseline) and 12 minutes after (response) test product intake
Changes from baseline in the BOLD signal | Six minutes before (baseline) and 12 minutes after (response) test product intake
  Using whole brain approach as well as seed based (hypothalamus, prefrontal cortex, nucleus accumbens, Ventral Tegmental Area, Amygdala).

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen van der Grond, Dr., Principal Investigator — Leiden University Medical Center
Locations (1):
- Leids Universitair Medisch Centrum, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lodi A, Zarantonello L, Bisiacchi PS, Cenci L, Paoli A. Ketonemia and Glycemia Affect Appetite Levels and Executive Functions in Overweight Females During Two Ketogenic Diets. Obesity (Silver Spring). 2020 Oct;28(10):1868-1877. doi: 10.1002/oby.22934. Epub 2020 Sep 1. PMID 32875733
- [Derived] Van Opstal AM, Hafkemeijer A, van den Berg-Huysmans AA, Hoeksma M, Mulder TPJ, Pijl H, Rombouts SARB, van der Grond J. Brain activity and connectivity changes in response to nutritive natural sugars, non-nutritive natural sugar replacements and artificial sweeteners. Nutr Neurosci. 2021 May;24(5):395-405. doi: 10.1080/1028415X.2019.1639306. Epub 2019 Jul 10. PMID 31288630